CLINICAL TRIAL: NCT05766423
Title: Phenotyping Adherence Through Technology-Enabled Reports and Navigation: The PATTERN Study
Brief Title: Phenotyping Adherence Through Technology-Enabled Reports and Navigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: The Claude D. Pepper Older Americans Independence Centers (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00217555; P30AG059988 (NIH)
Record Dates: First submitted 2023-02-17; First posted 2023-03-13 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care includes:
  1. The normal standard clinical practices at the participating practice.
  2. No specific materials to promote PATTERN, and no additional materials that include adherence assessments or care alert notifications.
- The PATTERN Intervention (Active Comparator): The intervention components include:
  1. An adherence assessment completed by participants ahead of a regularly scheduled clinic visit.
  2. Care alert notifications directed to a nurse pool and/or member of the clinical care team.
  Interventions: Behavioral: The PATTERN Intervention

INTERVENTIONS:
Behavioral: The PATTERN Intervention — The intervention components include:
  1. An adherence assessment that requests patients to self-report via MyChart about their medication use. The assessment provides a link between the health center and the patient ahead of a regularly scheduled clinic visit.
  2. Care alert notifications directed to a nurse pool and/or member of the clinical care team when a medication adherence related problem is identified by the adherence assessment. The alert will also include the type of problem the patient is experiencing (cognitive, psychological, medical, regiment, social and/or economic). Once they receive these alerts, the care team can then activate appropriate staff and/or resources to respond.
  Arms: The PATTERN Intervention

SUMMARY:
This study is being conducted to adapt and pilot test a technology-enabled, primary care strategy for routinely monitoring medication use and adherence among older adults with multiple chronic conditions and polypharmacy.

DETAILED DESCRIPTION:
Our study aims are to:

Aim 1: Adapt the PATTERN intervention for use in primary care using input from key stakeholders. During Aim 1, the Northwestern research team will solicit opinions from key informants (patients, clinicians, practice administrators) to ensure PATTERN meets the needs of primary care.

Aim 2: Assess the PATTERN intervention's feasibility and acceptability for use in primary care. During Aim 2, the investigators will conduct a 2-arm, patient-randomized controlled trial at a Northwestern Medicine primary care practice. Participants will be recruited and randomly assigned, using a random number generator application, to either the PATTERN intervention or usual care. Usual care refers to the normal standard clinical practices at the participating practice. Participants will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

Each participant must:

* Be an adult aged 65 or older
* Speak English as their primary language
* Have multiple chronic conditions
* Be prescribed 8 or more medications
* Be primarily responsible for administering own medication
* Receive medical care at the participating primary care practice
* Have access to the internet and an active email address
* Be signed up for the patient portal (MyChart)

Exclusion Criteria:

No participant can:

* Have severe, uncorrectable visual, hearing or cognitive impairments that would preclude study consent or participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Pack, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 539 assessed participants, 73 met inclusion criteria and were randomized and allocated to Usual Care(n=36) and Intervention group(n=37). Of 36 allocated in Usual Care, 1 participant withdrawn and 3 consented but didn't schedule an interview, therefore were excluded from the study. Of 37 allocated in Intervention group, 5 participants consented but did not schedule an interview, therefore were excluded from the study.
Groups:
- The PATTERN Intervention: The intervention components include:
  1. An adherence assessment completed by participants ahead of a regularly scheduled clinic visit.
  2. Care alert notifications directed to a nurse pool and/or member of the clinical care team.
  The PATTERN Intervention: The intervention components include:
  1. An adherence assessment that requests patients to self-report via MyChart about their medication use. The assessment provides a link between the health center and the patient ahead of a regularly scheduled clinic visit.
  2. Care alert notifications directed to a nurse pool and/or member of the clinical care team when a medication adherence related problem is identified by the adherence assessment. The alert will also include the type of problem the patient is experiencing (cognitive, psychological, medical, regiment, social and/or economic). Once they receive these alerts, the care team can then activate appropriate staff and/or resources to respond.
Period: Overall Study
Arm/Group | Usual Care | The PATTERN Intervention
Started | 36 | 37
Completed | 32 | 32
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Consented, not scheduled | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | The PATTERN Intervention | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (7.5) | 74.9 (6.1) | 75.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 12 | 10 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 1 participant in intervention group with missing race data.
  Participants
    Race: White | 19 | 18 | 37
    Race: Black or African American | 11 | 12 | 23
    Race: Asian Indian | 0 | 1 | 1
    Race: Japanese | 1 | 0 | 1
    Race: Other | 1 | 0 | 1
    Race: Refused | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 29 | 31 | 60
  Ethnicity: Hispanic or Latino | 1 | 0 | 1
  Ethnicity: Refused | 2 | 1 | 3
Health Status [Count of Participants; unit: Participants] — The participants were asked about their self-reported overall health. The measure is a 5-point Likert scale range from excellent health to poor health.
  Participants
    Excellent | 1 | 0 | 1
    Very good | 3 | 8 | 11
    Good | 17 | 12 | 29
    Fair | 10 | 10 | 20
    Poor | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: Participants' medication adherence will be measured at about 2-4 weeks after their clinic visit using a validated self-report measure: ASK-12. The 12-item measure assesses general medication attitudes and beliefs across three domains: 1) inconvenience/forgetfulness, 2) treatment beliefs, and 3) behaviors. Response options range from "Strongly Disagree" to "Strongly Agree". Scores can range from 12-60 with higher scores representing greater barriers to adherence.
Time Frame: About 2-4 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | The PATTERN Intervention
Number analyzed (Participants) | 32 | 32
score on a scale | 21.6 (6.2) | 23.8 (7.0)

2. Secondary Outcome: Fidelity
Description: The investigators will examine participants' completion rates of the routine medication adherence assessment. This will be identified via the EHR.
Time Frame: By the scheduled clinic visit (baseline)
Population: Only the participants in PATTERN Intervention group were sent the medication adherence assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | The PATTERN Intervention
Number analyzed (Participants) | 0 | 32
Participants | 0 | 15

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and nonserious adverse events were not assessed for the participants in this study.
Arm/Group | Usual Care | The PATTERN Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT05766423/Prot_000.pdf
  • Informed Consent Form (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT05766423/ICF_001.pdf